CLINICAL TRIAL: NCT06072183
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, 52-WEEK PLACEBO-CONTROLLED MULTI-CENTER STUDY WITH A DOUBLE-BLIND 52-WEEK EXTENSION PERIOD WITH RANDOMIZED DOSE UP/DOSE DOWN TITRATION INVESTIGATING THE EFFICACY, SAFETY, AND TOLERABILITY OF RITLECITINIB IN ADULT PARTICIPANTS WITH NONSEGMENTAL VITILIGO
Brief Title: A 104-Week Study of Ritlecitinib Oral Capsules in Adults With Nonsegmental Vitiligo (Active and Stable) Tranquillo 2
Acronym: Tranquillo 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981080; 2022-502518-98-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Stable Nonsegmental Vitiligo; Active Nonsegmental Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1- Ritlecitinib 100 milligrams (mg) (Experimental): Randomized to Ritlecitinib 100 mg QD for 52 weeks before progressing into the up/down titration extension period, rerandomized according to responder status.
  Interventions: Drug: Ritlecitinib
- Arm 2- Ritlecitinib 50mg (Experimental): Randomized to Ritlecitinib 50 mg QD for 52 weeks before progressing into the up/down titration extension period, rerandomized according to responder status.
  Interventions: Drug: Ritlecitinib
- Arm 3- Placebo (Placebo Comparator): Randomized to Placebo QD for 52 weeks before progressing into the up/down titration extension period, rerandomized according to responder status.
  Interventions: Drug: Placebo
- Arm 4- Ritlecitinib 100mg (Experimental): Non-randomized open-label Ritlecitinib 100mg QD for 52 weeks.
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — 100mg Capsule
  Arms: Arm 1- Ritlecitinib 100 milligrams (mg); Arm 4- Ritlecitinib 100mg
Drug: Ritlecitinib — 50mg Capsule
  Arms: Arm 2- Ritlecitinib 50mg
Drug: Placebo — Matching capsule
  Arms: Arm 3- Placebo

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine ritlecitinib for the possible treatment of nonsegmental vitiligo. Vitiligo causes white patches on your skin when the cells that give your skin color are destroyed. Nonsegmental means that it can affect both sides of the body such as both knees and both hands.

Ritlecitinib has been tested in earlier clinical studies and has a favorable safety profile. At present there are no approved medications taken by mouth to treat nonsegmental vitiligo.

This study is seeking participants who:

* Are 18 years of age or older.
* are confirmed to have nonsegmental vitiligo for at least 3 months.
* Are willing to stop all other treatments that they may be taking for vitiligo.

In this study participants will be chosen by chance, like drawing names out of a hat to receive 1 of 3 treatments:

•Part I where two different amounts of ritlecitinib (50 mg and 100 mg) are taken once daily. It will be compared to placebo. Placebo is a dummy capsule. It doesn't have any medicine used in the study.

Participants receiving placebo who have not responded to treatment after 52 weeks will be given 100 milligrams or 50 milligrams of ritlecitinib for the remaining 52 weeks of the study.

• In Part II, participants will only receive 100 milligrams of ritlecitinib. About 1000 participants will take part in Part I and around 450 in Part II globally. The study will compare the experiences of people receiving ritlecitinib to those of the people who do not. This will help see if ritlecitinib is safe and effective.

People in Part I will be in this study for about 26 months and people in Part II will be in this study for about 14 months. During the study, participants in part I will need to visit the study site at least 17 times. In part II, participants will visit at least 11 times.

Participants will undergo various tests and procedures such as:

* vitiligo rating,
* physical examinations,
* hearing tests,
* blood tests,
* x-ray,
* ECG,
* photographs of areas with vitiligo. Participants will be asked to complete questionnaires about their vitiligo.

DETAILED DESCRIPTION:
Study B7981080 is a Phase 3 randomized, double-blind, multicenter study with a 52-week placebo-controlled period (Part Ia) followed by a double-blind 52-week extension period (Part Ib) that includes randomized dose-up/down titration and a de novo 52-week non-randomized open-label cohort (Part II), investigating the efficacy, safety, and tolerability of ritlecitinib 100 mg QD and 50 mg QD compared with placebo in adult participants with nonsegmental active or stable vitiligo

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 years (or the minimum age of consent in accordance with local regulations) or older (no upper age limit) at Screening.

   • Meeting reproductive criteria for female participants.

   Disease Characteristics:
2. Eligible participants must have at both Screening and BL:

   * A clinical diagnosis of nonsegmental vitiligo for at least 3 months; and
   * BSA involvement 4% to 60% inclusive, excluding involvements at palms of the hands, soles of the feet, or dorsal aspect of the feet and
   * BSA ≥0.5% involvement on the face. Face is defined as including the area on the forehead to the original hairline, on the cheek to the jawline vertically to the jawline and laterally from the corner of the mouth to the tragus. Face will not include scalp, ears, neck, or surface area of the lips, but will include the nose and the eyelids; and
   * F-VASI ≥0.5 and T-VASI ≥3; and
   * Either active or stable nonsegmental vitiligo at Screening and BL visits. All participants who do not have the features of active vitiligo (defined below) will be classified as having stable disease.

   Active vitiligo is defined as:

   Participants will be classified as having active vitiligo based on the presence of at least one active lesion at BL defined as one of the following:
   * New/extending lesions(s) in the 3 months prior to Screening visit (confirmed by photographs or medical record);
   * Confetti-like lesion(s); Confetti-like depigmentation is characterized by the presence of numerous 1-mm to 5-mm depigmented macules in clusters;
   * Trichrome lesion(s); Trichrome lesions have a hypopigmented zone of varying width between normal and completely depigmented skin, resulting in 3 different hues of skin;
   * Koebner phenomenon/phenomena (excluding Type 1 [history based on isomorphic reaction]). The Koebner phenomenon manifests as depigmentation at sites of trauma, usually in a linear arrangement.

   Stable vitiligo is defined as:

   • Participants will be classified as having stable vitiligo based on an absence of signs of active disease. All participants who do not have the features of active vitiligo (defined above) will be classified as having stable disease.

   Eligibility is determined at Screening and Baseline based on the resulting scores from the local in-person reads of F-VASI, T-VASI, and BSA.
3. Additional inclusion criteria are:

   * If receiving concomitant medications for any reason other than vitiligo, participant must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1. Participant must be willing to stay on a stable regimen during the duration of the study.
   * Must agree to stop all other treatments for vitiligo from Screening through the final follow-up visit.

Exclusion Criteria:

Medical Conditions:

1. Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.

   • Any psychiatric condition including recent or active suicidal ideation or behavior that meets defined criteria.
2. Medical conditions pertaining to vitiligo and other diseases/conditions affecting the skin:

   * Participants that have other types of vitiligo that do not meet criteria for active or stable vitiligo as noted in inclusion criteria (including but not limited to segmental vitiligo and mixed vitiligo).
   * Currently have active forms of other hypopigmentation (including but not limited to Vogt-Koyanagi-Harada disease, malignancy-induced hypopigmentation [melanoma and mycosis fungoides], post-inflammatory hypopigmentation, pityriasis alba [minor manifestation of atopic dermatitis], senile leukoderma [age-related depigmentation], chemical/drug-induced leukoderma, ataxia telangiectasia, tuberous sclerosis, melasma, and congenital hypopigmentation disorder including piebaldism, Waardenburg syndrome, hypomelanosis of Ito, incontinentia pigmenti, dyschromatosis symmetrica hereditarian, xeroderma pigmentosum, and nevus depigmentosus). NOTE: Coexistence of halo nevus/nevi (also known as Sutton nevus/nevi) is permitted.
   * Currently have active forms of inflammatory skin disease(s) or evidence of skin conditions (for example, but not limited to morphea, discoid lupus, leprosy, syphilis, psoriasis, seborrheic dermatitis) at the time of the Screening or BL Visit that in the opinion of the investigator would interfere with evaluation of vitiligo or response to treatment.
   * Leukotrichia in more than 33% of the face surface area affected with vitiligo lesions or leukotrichia in more than 33% of the total body surface area affected with vitiligo lesions.
   * Have a superficial skin infection within 2 weeks prior to first dose on Day 1. NOTE: participants may be rescreened after the infection resolves.
3. General Infection History:

   * Have a history of systemic infection requiring hospitalization, parenteral antimicrobial, antiviral (including biologic treatment), antiparasitic, antiprotozoal, or antifungal therapy, or as otherwise judged clinically significant by the investigator within 6 months prior to Day 1.
   * Have active acute or chronic infection requiring treatment with oral antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to Day 1. NOTE: participants may be rescreened after the infection resolves.
   * Evidence or history of untreated, currently treated or inadequately treated active or latent infection with Mycobacterium tuberculosis.
4. Specific Viral Infection History:

   * History (single episode) of disseminated HZ or disseminated herpes simplex or recurrent (more than one episode of) localized, dermatomal HZ.
   * Infected with HBV or HCV: all participants will undergo screening for HBV and HBC for eligibility.
   * Participants who are positive for HCVAb and HCV RNA will not be eligible for this study.
   * Have a known immunodeficiency disorder (including positive serology for HIV at screening) or a first-degree relative with a hereditary immunodeficiency.
5. Other Medical Conditions:

   * Current or recent history of clinically significant severe, progressive, or uncontrolled renal (including but not limited to active renal disease or recent kidney stones), hepatic, hematological, gastrointestinal, metabolic, endocrine (eg, untreated hypovitaminosis D or hypothyroidism), pulmonary, cardiovascular, psychiatric, immunologic/rheumatologic or neurologic disease; or have any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or interfere with the interpretation of study results; or in the opinion of the investigator or Pfizer (or designee), the participant is inappropriate for entry into this study, or unwilling/unable to comply with study procedures and lifestyle requirements.
   * History of severe allergic or anaphylactoid reaction to any kinase inhibitor or a known allergy/hypersensitivity to any component (including excipients) of the study intervention.
   * Have hearing loss with progression over the previous 5 years, sudden hearing loss, or middle or inner ear disease such as otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered current, fluctuating, or progressive.
   * Have a history of any lymphoproliferative disorder such as EBV-related lymphoproliferative disorder, history of lymphoma, history of leukemia, or signs and symptoms suggestive of current lymphatic or lymphoid disease.
   * Abnormal findings on the Screening chest imaging (eg, chest x-ray). Chest imaging may be performed up to 12 weeks prior to screening. Documentation of the official reading must be located and available in the source documentation.
   * Long QT Syndrome, a family history of Long QT Syndrome, or a history of TdP.
   * Have any malignancies or have a history of malignancies with the exception of adequately treated or excised nonmetastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ.
   * Significant trauma or major surgery within 1 month of the first dose of study drug or considered in imminent need for surgery or with elective surgery scheduled to occur during the study.

   Prior/Concomitant Therapy:
6. Have received any of the prohibited treatment regimens specified.

   Prior/Concurrent Clinical Study Experience:
7. Previous administration with an investigational drug or vaccine that do not affect vitiligo within 4 weeks of Day 1 [Baseline] or within 5 half-lives, whichever is longer.

   Diagnostic Assessments:

   Any of the following abnormalities in clinical laboratory tests at Screening, as assessed by the study-specific laboratory and, if deemed necessary, confirmed by a single repeat:
8. Renal impairment
9. Hepatic dysfunction
10. Other laboratory abnormalities
11. Standard 12-lead ECG that demonstrates clinically relevant abnormalities

    Other Exclusion Criteria:
12. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1571 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
US only Co-Primary Endpoints: Response based on Facial Vitiligo Area Scoring Index 75 (F-VASI75) at Week 52 and Total body Vitiligo Area Scoring Index 50 (T-VASI50) at Week 52 | 52 Weeks
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline) and T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
Global (Other than US): Response based on Facial Vitiligo Area Scoring Index 75 (F-VASI75) at Week 52 | 52 Weeks
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline).
Incidence of Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events (AEs) leading to discontinuation. | Baseline through 108 weeks
  To evaluate the safety and tolerability of ritlecitinib in adult participants with non segmental vitiligo
Incidence of Clinically significant laboratory abnormalities. | Baseline through 108 weeks

SECONDARY OUTCOMES:
Response based on F-VASI75 at 24 and 36 weeks | 24 and 36 Weeks
  Proportion of participants achieving at least a 75% improvement in F-VASI from Baseline.
US-Only: Response based on T-VASI50 at 24 and 36 weeks | 24 and 36 weeks
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline).
Global (Other than US):Patient Global Impression of Severity-Face (PGIS-F) | Week 24, 36 and week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIS-F at Week 24, 36 and 52
Global (Other than US): Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) | Week 24, 36 and week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIS-V at Week 24, 36 and 52
Global (Other Than US): Response based on T-VASI50 at Week 24, 36 and 52 | Week 24, 36 and 52
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline).
Patient Global Impression of Change-Face (PGIC-F) | Week 36 and week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-F at Weeks 36 and 52.
Patient Global Impression of Change- Overall vitiligo(PGIC-V) | Week 36 and week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIC-V at Weeks 36 and 52.
Change from baseline in Dermatology Life Quality Index (DLQI) | Week 52
  To evaluate the change from baseline in DLQI at week 52
Proportion of participants achieving disease stabilization | Baseline through week 104
  The difference in the proportion of participants with stable disease at all timepoints in participants with non segmental vitiligo treated with ritlecitinib 50 mg QD and 100mg compared to placebo
Response based on T-VASI50 | Baseline through week 4, week 8, week 12, week 48, week 56, week 60, week 64, week 76, week 88 and week 104.
  Proportion of participants achieving T-VASI50 (defined as at least 50% improvement in T-VASI from Baseline)
Response based on F-VASI75 | Baseline through week 4, week 8, week 12, week 48, week 56, week 60, week 64, week 76, week 88 and week 104.
  Proportion of participants achieving F-VASI75 (defined as at least 75% improvement in F-VASI from Baseline)
Response based on T-VASI75 | Baseline through week 4, week 8, week 12, week 24, week 36, week 48, week 56, week 60, week 64, week 76, week 88 and week 104.
  Proportion of participants achieving T-VASI75 (defined as at least 75% improvement in T-VASI from Baseline)
Global (Other than US): Response based on T-VASI75 | Baseline through week 52
  Proportion of participants achieving T-VASI75 (defined as at least 75% improvement in T-VASI from Baseline)
Proportion of participants with sustained improvement in T-VASI | Week 36 through week 52
  Defined as maintenance of ≥T-VASI50 from Week 36 to Week 52
Proportion of participants with sustained improvement in F-VASI | Week 36 through week 52
  Defined as maintenance of ≥F-VASI75 from Week 36 to 52
Time to rescue medication use | Baseline through week 104
US-Only: Percentage change from baseline (% CFB) in F-VASI at Weeks 24, 36 and 52 | Weeks 24, 36 and 52
  To compare the efficacy of ritlecitinib 100 mg QD versus placebo on % CFB in F-VASI at Weeks 24, 36 and 52
US-Only: % CFB in T-VASI at weeks 24, 36 and 52 | Weeks 24, 36 and 52
  To compare the efficacy of ritlecitinib 100 mg QD versus placebo on % CFB in T-VASI at Weeks 24,36 and 52
Response based on T-VASI90 | Baseline through week 52
  Proportion of participants achieving T-VASI90 (defined as at least 90% improvement in T-VASI from Baseline)
Response based on T-VASI100 | Baseline through week 52
  Proportion of participants achieving T-VASI90 (defined as at least 100% improvement in T-VASI from Baseline)
Response based on F-VASI50 | Baseline through week 104
  Proportion of participants achieving F-VASI50 (defined as at least 50% improvement in F-VASI from Baseline).
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) | Week 52
  To assess the effect of ritlecitinib compared to placebo on depression and anxiety subscales of the HADS at week 52
The proportion of patients achieving absence of depression on HADS depression subscale | Week 52
  Response based on a 'normal' subscale score indicative of an absence of depression (in participants with baseline HADS subscale scores indicative of depression)
The proportion of patients achieving absence of anxiety on HADS anxiety subscale | Week 52
  Response based on a 'normal' subscale score indicative of an absence of anxiety (in participants with baseline HADS subscale scores indicative of anxiety)
US-Only: Patient Global Impression of Severity-Face (PGIS-F) | Week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIS-F at 52
US-Only: Patient Global Impression of Severity-Overall Vitiligo (PGIS-V) | Week 52
  To assess the effect of ritlecitinib compared to placebo on the PGIS-V at 52
% CFB in F-VASI at Week 4, 8, 12, 48, 56, 60, 64, 76, 88 and 104. | Baseline through week 104
  To compare the efficacy of ritlecitinib 100 mg QD versus placebo on % CFB in F-VASI at all time points
% CFB in T-VASI at Week 4, 8, 12, 48, 56, 60, 64, 76, 88 and 104. | Baseline through week 104
  To compare the efficacy of ritlecitinib 100 mg QD versus placebo on % CFB in T-VASI at all time points

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (229):
- United States (67):
  - Center for Dermatology and Plastic Surgery/CCT Research, Scottsdale, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - First OC Dermatology Research Inc, Fountain Valley, California
  - Seaside Audiology Vertigo & Ear Specialists, Huntington Beach, California
  - Wallace Medical Group, Inc, Los Angeles, California
  - Kaiser Permanente, Oakland, California
  - Cura Clinical Research - Oxnard, Oxnard, California
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Integrative Skin Science and Research, Sacramento, California
  - University of California San Diego - La Jolla, San Diego, California
  - Wolverine Clinical Trials, Santa Ana, California
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - FXM Clinical Research - Fort Lauderdale, Fort Lauderdale, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Harmony Medical Research Institute, Hialeah, Florida
  - Clever Medical Research, Miami, Florida
  - JD Medical Group, Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - SouthCoast Research Center, Miami, Florida
  - University of Miami, Miami, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - South Miami Medical & Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Skin Research of South Florida, Miami, Florida
  - Well Pharma Medical Research, Corp., Miami, Florida
  - FXM Clinical Research - Miami, Miami, Florida
  - Health and Life Research Institute, Miami, Florida
  - University of Miami, Kendall Office, Miami, Florida
  - Floridian Research Institute Llc, Miami, Florida
  - Sanitas Research, Miami, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - FXM Clinical Research - Miramar, Miramar, Florida
  - GCP Research, Global Clinical professionals, St. Petersburg, Florida
  - Advanced Clinical Research Institute, Tampa, Florida
  - USF Health, Tampa, Florida
  - Sidney P. Smith, MD, PC dba Georgia Skin & Cancer Clinic, Savannah, Georgia
  - NorthShore University Health System, Skokie, Illinois
  - Indiana University School of Medicine - Indiana CTSI Clinical Research Center, Indianapolis, Indiana
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The South Bend Clinic, LLC, South Bend, Indiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - CS Mott Center, Detroit, Michigan
  - Wayne Health, Detroit, Michigan
  - Henry Ford Medical Center - New Center One, Detroit, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - OptiSkin Medical, New York, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Darst Dermatology, Charlotte, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Columbia Dermatology & Aesthetics, Columbia, South Carolina
  - Palmetto Clinical Trial Services - Greenville, Greenville, South Carolina
  - Center for Clinical Studies, Houston, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Complete Dermatology, Sugar Land, Texas
  - The Woodlands Dermatology Associates, PA, The Woodlands, Texas
  - University of Utah, Murray, Utah
  - Springville Dermatology - Springville/CCT Research, Springville, Utah
  - The Education & Research Foundation, Inc., Forest, Virginia
- Australia (12):
  - Paratus Clinical Research Woden, Phillip, Australian Capital Territory
  - St George Dermatology & Skin Cancer Centre, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Veracity Clinical Research, Woolloongabba, Queensland
  - North Eastern Health Specialists, Campbelltown, South Australia
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Dr Rodney Sinclair Pty Ltd, East Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Institute for Skin, Health and Immunity, Mitcham, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
- Belgium (5):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-capitale, Région de
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-capitale, Région de
  - UZ Gent, Ghent, Oost-vlaanderen
  - UZ Leuven, Leuven, Vlaams-brabant
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Bulgaria (13):
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia (stolitsa)
  - Diagnostic Consultative Centre (DCC) - Foкus 5, Sofia, Sofia (stolitsa)
  - Clinic EvroDerma, Sofia, Sofia (stolitsa)
  - MHAT Pazardzhik, Pazardzhik
  - Diagnostic Consultative Center 1 - Pernik, Pernik
  - Medical Center Exacta Medica, Pleven
  - Medical Center Prolet EOOD, Rousse
  - Diagnostic Consultative Center "Ascendent", Sofia
  - Diagnostic - Consultative Center XXVIII - Sofia, Sofia
  - "Diagnostic - Consultative Center XX - Sofia" EOOD, Sofia
  - UMHAT "Prof. Dr. Stoyan Kirkovich"AD, Stara Zagora
  - Center for Skin and Venereal Diseases - Veliko Tarnovo, Veliko Tarnovo
  - Multiprofile Hospital for Active Treatment Sv. Panteleymon - Yambol AD, Yambol
- Canada (23):
  - Dermatology Research Institute, Calgary, Alberta
  - Alberta Dermasurgery Centre, Edmonton, Alberta
  - The Skin Care Centre, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - DermEffects, London, Ontario
  - DermEdge Research, Mississauga, Ontario
  - The Centre for Clinical Trials, Oakville, Ontario
  - JRB Research Inc., Ottawa, Ontario
  - York Dermatology Clinic & Research Centre, Richmond Hill, Ontario
  - North York Research Inc, Toronto, Ontario
  - Dermatology on Bloor - Research Toronto, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Montreal, Quebec
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Saint-Louis, Sherbrooke, Quebec
  - Diex Recherche Sherbrooke, Sherbrooke, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan
  - Saskatoon Dermatology Centre, Saskatoon, Saskatchewan
  - Diex Recherche Quebec, Québec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
  - Alpha Recherche Clinique, Québec
- China (22):
  - Beijing Friendship Hospital Affiliate of Capital University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - NanYang First people's hospital, Nanyang, Henan
  - The First Hospital of Wuhan, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Chengdu second people's hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shanghai General Hospital, Shanghai
- Germany (12):
  - Rosenpark Research GmbH, Darmstadt, Hesse
  - Klinikum Bielefeld gem. GmbH, Bielefeld, North Rhine-Westphalia
  - Klinikum Bielefeld Rosenhöhe, Bielefeld, North Rhine-Westphalia
  - Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Hautarztpraxis Dr. Gerlach, Dresden, Saxony
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden, Saxony
  - Hautarztpraxis Dr. Neubauer, Leipzig, Saxony
  - HNO-Praxis Dr. Kugler in Magdeburg, Magdeburg, Saxony-Anhalt
  - Magdeburger Company for Medical Studies and Services, Magdeburg, Saxony-Anhalt
  - Radiologie Ulrichshaus, Magdeburg, Saxony-Anhalt
- Hungary (8):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Synexus Magyarorszag Kft. (Gyula DRS), Gyula, Bekes County
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Óbudai Egészségügyi Centrum, Budapest
  - Orvostudomanyi Kutato es Fejleszto Kft, Debrecen
  - DERMA-B Egészségügyi és Szolgáltató, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Derm-Surg Kft., Kaposvár
- Italy (7):
  - ASL1 Avezzano-Sulmona-L'Aquila, L’Aquila, Abruzzo
  - Presidio Ospedaliero Firenze Centro Piero Palagi, Florence, Firenze
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - IRCCS Istituti Fisioterapici Ospitalieri, Roma, RM
  - Ospedale Israelitico, Rome, ROMA
  - Istituto Dermopatico Immacolata, Rome, ROMA
  - Ospedale Civile - Azienda Ospedaliera Universitaria di Cagliari, Cagliari
- Japan (10):
  - Japan Community Health Care Organization Chukyo Hospital, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Juntendo University Urayasu Hospital, Urayasu, Chiba
  - Takarazuka City Hospital, Takarazuka, Hyōgo
  - Tokyo Medical University Ibaraki Medical Center, Inashiki-gun, Ibaraki
  - Kindai University Nara Hospital, Ikoma, Nara
  - Osaka Habikino Medical Center, Habikino, Osaka
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Institute of Science Tokyo Hospital, Bunkyo-ku, Tokyo
  - Yamaguchi University Hospital, Ube, Yamaguchi
- Mexico (6):
  - Trials in Medicine, Mexico City, Mexico City
  - Clinica de Enfermedades Cronicas y Procedimientos Especiales, SC, Morelia, Michoacán
  - Centro Regiomontano de Investigación, Monterrey, Nuevo León
  - Servicios Hospitalarios de Mexico S.A. DE C.V., Chihuahua City
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Arké SMO S.A de C.V, Veracruz
- Poland (11):
  - Clinica Dermatoestetica Prywatny Gabinet Dermatologiczny I Alergologiczny Prof.Dr Hab.Med. Barbara Z, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy, Marek Brzewski, Paweł Brzewski spółka, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne, Krakow, Lesser Poland Voivodeship
  - ETG Warszawa, Warsaw, Masovian Voivodeship
  - Klinika Ambroziak Dermatologia, Warsaw, Masovian Voivodeship
  - Royalderm Agnieszka Nawrocka, Warsaw, Masovian Voivodeship
  - Specderm Poznanska sp.j., Bialystok, Podlaskie Voivodeship
  - ClinicMed Daniluk, Nowak Spółka komandytowa, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Twoja Przychodnia SCM, Szczecin, West Pomeranian Voivodeship
  - "DERMED" Centrum Medyczne Sp. z o.o., Lodz, Łódź Voivodeship
- Puerto Rico (3):
  - Cardiovascular Radiology Institute, San Juan
  - Clinical Research Puerto Rico, San Juan
  - Centro de Audiología y Balance, San Juan
- Slovakia (8):
  - Fakultna nemocnica s poliklinikou F.D.Roosevelta Banska Bystrica, Banská Bystrica, Banská Bystrica Region
  - SANARE, s.r.o, Svidník, Presov
  - Fakultna nemocnica Trnava, Trnava, Trnava Region
  - CLINIQ s.r.o., Bratislava
  - BeneDerma, Bratislava
  - Derma therapy spol. s.r.o., Bratislava
  - Topskin pro s.r.o., Košice
  - Poliklinika ProCare Kosice s.r.o., Košice
- Spain (13):
  - AUDIKA, Córdoba, Andalusia
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Germans Trias i Pujol, Badalona, Barcelona [barcelona]
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona [barcelona]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [cataluña]
  - Clínica Gaias - Santiago, Santiago de Compostela, Galicia [galicia]
  - Hospital Universitario Infanta Leonor, Madrid, Madrid, Comunidad de
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínica Gaias - Santiago, Santiago de Compostela
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (5):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (2):
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Bezmialem Vakf Üniversitesi, Istanbul
- United Kingdom (2):
  - West Middlesex University Hospital, Isleworth, England
  - Guy's & St Thomas' NHS Foundation Trust, London, London, CITY of

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981080